CLINICAL TRIAL: NCT03684239
Title: The Effect of G-CBT on the Patients With AN : A Randomized Controlled Trial
Brief Title: The Effect of G-CBT on the Patients With AN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Jue CHEN, Director of Psychosomatic Department in Shanghai Mental Health Center, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16411965200
Record Dates: First submitted 2018-09-23; First posted 2018-09-25 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Feeding and Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-CBT group (Experimental): G-CBT group has 40 patients, maybe will be divided them into 4 groups. Every group has 8-10 patients. Every group receive 10 times CBT group therapy and 1 times a week for 120 minutes each time.
  Interventions: Behavioral: G-CBT; Other: Conventional treatment
- Conventional treatment group (Active Comparator): Conventional treatment group has 40 patients, received routine outpatient treatment. Once every two weeks for 45 minutes each time, including nutritional advice, encouragement, and routine treatment by a psychiatrist with work experience with eating disorders.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Behavioral: G-CBT — CBT is based on the model that there is a interaction between cognition, emotion and behavior. The way people think affects the way they feel and the behavior they do. And then the feelings in turn affect how they think,So it is valid for AN patient.
  Arms: G-CBT group
Other: Conventional treatment — Conventional treatment including nutritional advice, encouragement, and routine treatment by a psychiatrist with work experience with eating disorders.

SUMMARY:
The study is to examine whether the G-CBT for anorexia nervosa is effective or not. The study will use randomized controlled study design. 80 patients with AN will be recruited from Shanghai Mental Health Center, There will be two groups: CBT treatment group and conventional treatment group. Each group is 40 and then the CBT group will be given standard CBT intervention for 12 weeks. The control group will receive outpatient treatment. To assess the eating disorder symptoms, impulsive and emotional change, clinical symptom scales, psychological scales and the security indexs will be used at baseline, 4 weeks, 8 weeks, 12 weeks (end of treatment), 24 weeks (3 months after treatment) and 36 weeks (6 months after treatment follow-up).

DETAILED DESCRIPTION:
Eating disorder is a chronic mental disorder characteristic of abnormal eating behaviors and psychological disorders, accompanied by significant weight changes and physiological dysfunction. Many people with EDs have cognitive disorder of their body shape or body weight. Anorexia is a subtype of EDs. The main feature of anorexia nervosa is the extreme attention to body weight and body shape. As a result of this conflict the patients could be malnutrition, metabolism and endocrine disorders with significant weight loss. And women may have amenorrhea. At the mean time, the patient will also have a lot of mental symptoms such as depression, anxiety and obsession.

The disease mostly occurs in adolescents and young women. The prevalence rates in Europe and America is 0.5%-3.7%, 90% of which are women. The course of the disease is chronic, the average duration of disease is 4-6 years. Furthermore the mortality rate is high, a 20-year follow-up data shows that the mortality rate is nearly 20%. Most of the causes of death are physical complications and depression.

However, due to the special psychological behavior mechanism, patients have almost no willingness to be treated. As well as the long duration of disease and the highrisk of drug therapy, it all causes the great difficulties in the treatment. Many patients may even suffer from eating disorders for a lifetime. On another hand, the effective treatment options are still inconclusive. Psychotherapy, especially and cognitive behavior, is one of the most effective treatments at present.

On the other hand, psychotherapy is quite expensive, requiring not only a large number of qualified therapists, but also a long treatment time. Which leads to a high treatment cost. In order to reduce the cost of treatment, group therapy is a reasonable choice. However, currently there are no related research reports in china.

Our study is to examine whether the G-CBT for anorexia nervosa is effective or not. The study will use randomized controlled study design. 80 patients with AN will be recruited from Shanghai Mental Health Center, There will be two groups: CBT treatment group and conventional treatment group. Each group is 40 and then the CBT group will be given standard CBT intervention for 12 weeks. The control group will receive outpatient treatment. To assess the eating disorder symptoms, impulsive and emotional change, clinical symptom scales, psychological scales and the security indexs will be used at baseline, 4 weeks, 8 weeks, 12 weeks (end of treatment), 24 weeks (3 months after treatment) and 36 weeks (6 months after treatment follow-up).

This study was designed with sufficient consideration about innovation as well as feasibility, and is to be operated on well proved theoretical basis and guidance of an operation manual. If successful, results of this study may bring great improvement to clinical practice of this refractory mental disorder.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14-30 years;
* right handedness;
* above primary education;
* met DSM-V criteria for AN

Exclusion Criteria:

* diagnosed with a mental illness;
* with severe physical or cognitive impairment

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Examination Questionnaire(EDE-Q) | Change from Baseline eating attitudes and behaviors at 4 weeks,8weeks,12weeks,24weeks,36weeks.
  Eating Disorder Examination Questionnaire can evaluate the eating disorder behavior and psychology characteristics and assess their frequency and intensity, which can assess the severity of eating disorders.It is a 41 item self-report questionnaire. It retains the format of the EDE including the 4 subscales (1. Restraint; 2. Eating concern; 3. Shape concern; 4. Weight concern) and global score. It also concerns behaviors over a 28-day time period and retains the scoring system of 0-6, with 0 indicating no days, 1=1-5 days, 2=6-12 days, 3=13-15 days, 4=16-22 days, 5=23-27 days and 6= every day.The scoring method is the sum of the scores for each item divided by the number of items.

SECONDARY OUTCOMES:
Eating Disorder Inventory(EDI) | Change from Baseline eating attitudes and behaviors at 12weeks,24weeks,36weeks.
  EDI can assess the eating attitudes and behaviors. It can evaluate the pathologic psychological characteristics of AN patients.comprises 64 questions, divided into eight subscales. Each question is on a 6-point scale (ranging from 'always' to 'never'), rated 0-3. The score for each sub-scale is then summed. There are 8 subscale scores on the EDI
Beck Depression Inventory（BDI-II） | Change from Baseline eating attitudes and behaviors at 4 weeks,8weeks,12weeks,24weeks,36weeks.
  Measurement of the severity of the symptoms of depression. It is consisted of twenty-one questions about how the subject has been feeling in the last week. Each question had a set of at least four possible responses, ranging in intensity. When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. Higher total scores indicate more severe depressive symptoms.
Beck Anxiety Inventory（BAI） | Change from Baseline eating attitudes and behaviors at 4 weeks,8weeks,12weeks,24weeks,36weeks.
  Measurement of the severity of the symptoms of anxiety.The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jue Chen, PHD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and baseline characteristics of participants
Supporting Information: Study Protocol, SAP
Time Frame: when the investigators ended the experiment at 2019, the investigators will share the data.
Access Criteria: CBT;Cognitive Behavioral Group Therapy; AN; Anorexia Nervosa

REFERENCES:
- [Background] Wonderlich S, Mitchell JE, Crosby RD, Myers TC, Kadlec K, Lahaise K, Swan-Kremeier L, Dokken J, Lange M, Dinkel J, Jorgensen M, Schander L. Minimizing and treating chronicity in the eating disorders: a clinical overview. Int J Eat Disord. 2012 May;45(4):467-75. doi: 10.1002/eat.20978. Epub 2012 Jan 23. PMID 22271525
- [Background] Groff SE. Is enhanced cognitive behavioral therapy an effective intervention in eating disorders? A review. J Evid Inf Soc Work. 2015;12(3):272-88. doi: 10.1080/15433714.2013.835756. Epub 2015 Jan 30. PMID 25661898
- [Background] Brown TA, Keel PK. Current and emerging directions in the treatment of eating disorders. Subst Abuse. 2012;6:33-61. doi: 10.4137/SART.S7864. Epub 2012 Mar 29. PMID 22879753
- [Background] Costa MB, Melnik T. Effectiveness of psychosocial interventions in eating disorders: an overview of Cochrane systematic reviews. Einstein (Sao Paulo). 2016 Apr-Jun;14(2):235-77. doi: 10.1590/S1679-45082016RW3120. PMID 27462898
- [Background] de Zwaan M, Hilbert A, Swan-Kremeier L, Simonich H, Lancaster K, Howell LM, Monson T, Crosby RD, Mitchell JE. Comprehensive interview assessment of eating behavior 18-35 months after gastric bypass surgery for morbid obesity. Surg Obes Relat Dis. 2010 Jan-Feb;6(1):79-85. doi: 10.1016/j.soard.2009.08.011. Epub 2009 Sep 3. PMID 19837012
- [Background] Fairburn CG, Cooper Z, Doll HA, O'Connor ME, Palmer RL, Dalle Grave R. Enhanced cognitive behaviour therapy for adults with anorexia nervosa: a UK-Italy study. Behav Res Ther. 2013 Jan;51(1):R2-8. doi: 10.1016/j.brat.2012.09.010. Epub 2012 Oct 22. PMID 23084515
- [Background] Watson HJ, Allen K, Fursland A, Byrne SM, Nathan PR. Does enhanced cognitive behaviour therapy for eating disorders improve quality of life? Eur Eat Disord Rev. 2012 Sep;20(5):393-9. doi: 10.1002/erv.2186. Epub 2012 Jun 22. PMID 22730260
- [Background] Dalle Grave R, El Ghoch M, Sartirana M, Calugi S. Cognitive Behavioral Therapy for Anorexia Nervosa: An Update. Curr Psychiatry Rep. 2016 Jan;18(1):2. doi: 10.1007/s11920-015-0643-4. PMID 26689208
- [Background] Polnay A, James VA, Hodges L, Murray GD, Munro C, Lawrie SM. Group therapy for people with bulimia nervosa: systematic review and meta-analysis. Psychol Med. 2014 Aug;44(11):2241-54. doi: 10.1017/S0033291713002791. Epub 2013 Nov 15. PMID 24238470
- [Derived] Gu L, Zou Y, Huang Y, Liu Q, Chen H, Chen J. The effect of group cognitive behavior therapy on Chinese patients with anorexia nervosa: an open label trial. J Eat Disord. 2021 Sep 15;9(1):114. doi: 10.1186/s40337-021-00469-7. PMID 34526151